CLINICAL TRIAL: NCT00362947
Title: Randomized Clinical Study of Different Treatment Doses and Duration of Low Molecular Weight Heparin (Parnaparin) in Superficial Vein Thrombosis
Brief Title: Different Doses and Duration of Low Molecular Weight Heparin (Parnaparin)in Superficial Vein Thrombosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, GUALTIERO PALARETI, Prof.Gualtiero Palareti, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: The Steflux study
Record Dates: First submitted 2006-08-11; First posted 2006-08-15 (Estimated); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Thrombophlebitis
Keywords: Superficial vein thrombosis; thrombophlebitis; LMWH; parnaparin
MeSH Terms: conditions — Thrombophlebitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A (Placebo Comparator): A - Parnaparin 8.500 UI aXa od (therapeutic doses) for 10 days followed by placebo for 20 days
  Interventions: Drug: LMWH parnaparin subcutaneously
- B (Active Comparator): B - Parnaparin 8.500 UI aXa od for 10 days followed by 6.400 UI aXa once daily (intermediate therapeutic doses) for 20 days
  Interventions: Drug: LMWH parnaparin subcutaneously
- C (Active Comparator): C - Parnaparin 4.250 UI aXa od (prophylactic doses) for 30 days
  Interventions: Drug: LMWH parnaparin subcutaneously

INTERVENTIONS:
Drug: LMWH parnaparin subcutaneously

SUMMARY:
The optimal treatment of superficial venous thrombosis (SVT) is still uncertain. Though low molecular weight heparin (LMWH) is considered the treatment of choice, studies conducted so far do not give clear indications of the optimal dose and duration of treatment. This study aims to evaluate whether an intermediate therapeutic dose of LMWH (parnaparin) is more effective than a prophylactic dose and also to assess whether 10 rather than 30 days are sufficient for treatment.

DETAILED DESCRIPTION:
Outpatients with an episode of SVT of the grand saphenous vein (for at least 4 cm), and/or SVT of the small saphenous vein (for at least 4 cm), and/or SVT of a collateral vein of the large saphenous vein of the thigh (for at least 4cm) are included in this prospective, randomised, double blind, national multicentre study.

Patients will be randomised into double-blind groups to receive (syringes will be identical in appearance) in consecutively numbered boxes:

A - Parnaparin, dose of 8,500 IU aXa taken subcutaneously once a day for 10 days B - Parnaparin, dose of 8,500 IU aXa per day for 10 days followed by Parnaparin 6,400 IU aXa per day for the subsequent three weeks. C - Parnaparin, dose of 4,250 IU aXa per day for 30 days Elastic compression treatment will be recommended with special stocking and/or elastic bandaging with compression to the ankles of 20-40 mmHg, where not contraindicated.

ELIGIBILITY:
Inclusion Criteria:

* Weight > 50 kg and less than 110 kg
* SVT of the grand saphenous vein for at least 4 cm
* SVT of the small saphenous vein for at least 4 cm
* Collateral SVT of the large saphenous vein of the thigh for at least 4cm

Exclusion Criteria:

* SVT of the grand saphenous vein reaching the saphenofemoral cross (within 3 cm)
* SVT of the small saphenous vein reaching the saphenopopliteal cross
* Documented proximal or distal DVT or pulmonary embolism
* SVT secondary to sclerotherapy
* Pregnancy and puerperium
* uncontrolled arterial hypertension (Systolic pressure > 180 mmHg and diastolic pressure > 110 mmHg)
* Active peptic ulcer
* Bacterial endocarditis
* Stroke in the previous 3 months
* Haemorrhagic diathesis
* Thrombocytopenia (platelets < 100,000/ µL)
* Hypersensitivity to heparin or history of thrombocytopenia induced by heparin
* Creatinine > 2 mg% (> 180 µmol/L)
* Heparin therapy (any dose) or anticoagulant therapy for longer than the previous 72 hours
* In-hospital development of SVT
* Previous saphenectomy by any method
* Surgery in the previous 30 days
* Serious liver disease
* Use of dextran, mannitol, thrombolytic treatment, chronic use of NSAID and cortisone-based drugs.
* Active cancer or under chemotherapy or radiotherapy
* Thrombectomy of superficial vein involved
* Refusal to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 664 (Actual)
Dates: Start 2006-08; Primary Completion 2010-09 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Primary effectiveness objectives | 33 days
  composite of symptomatic and asymptomatic DVT, relapse and/or symptomatic or asymptomatic local extension of SVT and symptomatic PE at 33 days.
Major bleeding | 33
  Bleeding events were defined as major if retroperitoneal, intracranial, intraocular with severe vision damage, intra-articular, intra-abdominal of upper or lower digestive tract, genito-urinary tract, respiratory tract or associated with a decrease in the haemoglobin of ≥ 2.0 g/dL, or if requiring transfusion of ≥2 units of blood or if fatal.
  Bleeding was classified as minor in all other cases.

SECONDARY OUTCOMES:
Secondary effectiveness objectives | 93
  i)- reduction in local symptoms during treatment and ii)- the combined efficacy end-point during a follow-up of 93 days after the start of treatment.
secondary outcome for safety | 33
  the composite of minor haemorrhages, thrombocytopenia or any other adverse events (e.g. local allergic reactions).

CONTACTS AND LOCATIONS:
Overall Officials: Gualtiero Palareti, MD, Study Chair — University of Bologna; Benilde Cosmi, MD PhD, Principal Investigator — University of Bologna
Locations (2):
- Italy (2):
  - Dept. Angiology & Blood Coagulation; University Hospital S.Orsola-Malpighi, Bologna, BO
  - U.O. Medicina Critica, Piacenza, PC

IPD SHARING:
Plan to Share IPD: No